CLINICAL TRIAL: NCT02630238
Title: The Effect of Branched-Chain Amino Acid Supplementation and Exercise on Body Composition During Energy Restriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor & Weider Research Chair Director, Exercise Nutrition Research Laboratory, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 10009692
Record Dates: First submitted 2015-12-09; First posted 2015-12-15 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Weight Loss; Obesity
Keywords: Exercise; Amino Acids, Branched-Chain
MeSH Terms: conditions — Weight Loss; Obesity; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Branched-Chain Amino Acid group (Experimental): The branched-chain amino acid group will be on a hypocaloric diet, exercise and receive 0.342g/kg of BCAA per day, partially accounted for through their diet with the rest provided by a BCAA supplement
  Interventions: Dietary Supplement: Branched-Chain Amino Acid Supplementation; Other: Exercise; Other: Diet
- Placebo Group (Placebo Comparator): The placebo will be on a hypocaloric diet, exercise and receive isoenergetic beverage with carbohydrate instead of branched-chain amino acids
  Interventions: Other: Placebo; Other: Exercise; Other: Diet

INTERVENTIONS:
Dietary Supplement: Branched-Chain Amino Acid Supplementation — All participants will partake in the same diet & exercise regime but this group will also be placed on a BCAA intake level of 0.342g/kg of BCAA per day
  Arms: Branched-Chain Amino Acid group
Other: Placebo — All participants will partake in the same diet & exercise regime but this group will receive an isocaloric placebo in form of carbohydrate solution
  Arms: Placebo Group
Other: Exercise — Exercise will take place in a class based, circuit training setting run by a certified personal trainer composed of both aerobic and lifting exercises
Other: Diet — Each participants will be placed on a daily energy deficit of 500 calories for the 8 week study period.

SUMMARY:
This double blind placebo study will take place over an 8 week treatment period of diet and exercise. All participants (n=16), in two groups, will be placed on the same hypocaloric diet and exercise program. Participants will be matched into pairs based on body fat % and then assigned into a test group & a placebo group. The placebo will be in the form of a powdered isoenergetic beverage with carbohydrate similar in taste & appearance to the powder BCAA supplement that the test group will receive. The test group will be put on 0.342g/kg of BCAA per day, partially accounted for through their diet with the rest provided by a BCAA supplement. At baseline, 4 weeks and 8 weeks habitual 3 day food logs, waist to hip ratio and BodPod measures of body fat & lean mass (both percentage & absolute values) will be taken for all participants.

DETAILED DESCRIPTION:
This double blind placebo study will take place over an 8 week treatment period of diet and exercise. All participants (n=16) will be placed on the same hypocaloric diet and exercise program. Both groups will exercise at the same time. Baseline habitual 3 day food logs, waist to hip ratio and BodPod measures of body fat & lean mass (both percentage & absolute values) will be taken for all participants. Each will be provided with macronutrient guidelines to follow (40% carbohydrate, 30% protein, 30% fat) & placed on a daily energy deficit of 500 calories for the 8 week study period. Participants in both treatment and control groups will be asked to record their dietary intake using the MyFitnessPal smartphone application or website in order to insure compliance to the prescribed diet. MyFitnessPal is a fast and easy to use calorie counter for Windows or phones. Further, it has the largest food database of any calorie counter apps (over 3,000,000 foods). Each individual will provide the investigators with a weekly screen shot of their mean data. Exercise will take place in a class based, circuit training setting run by a certified personal trainer (Alicia MacDougall). Exercise safety will be assessed by a Physical Readiness Questionnaire (the Par- Q and You - see appendix). Further, it is important to note that these women are overweight, not obese, and that research evidence indicates clearly that inactivity is far more hazardous to one's health than regular exercise (American College of Sports Medicine). Attendance will be recorded to document adherence. This style of training was chosen in order to combine both strength and endurance based training in an attempt to generate fat loss while keeping the workouts controlled by study investigators. Participants will be matched into pairs based on body fat % and then assigned into a test group & a placebo group. This ensures the groups will have similar mean and SD for fat mass at baseline. The placebo group will follow the diet and exercise regime described above plus, be given an isoenergetic placebo to take daily. The placebo will be in the form of a powdered isoenergetic beverage with carbohydrate instead of amino acids, similar in taste & appearance to the powder BCAA supplement that the test group will receive in order to keep the participants blind to their treatment. Specifically, the test group 0.342g/kg of BCAA per day, partially accounted for through their diet with the rest provided by a BCAA supplement (NOW BCAA Powder). The supplement will provide a 2:1:1 ratio of leucine, isoleucine, & valine respectively. At 4 and 8 week of treatment, all participants will be remeasured for waist to hip ratio and BodPod measures of body fat & lean mass. These values can then be compared to the baseline values for each of the study groups in order to determine if the increased BCAA intake proved to be effective. The beverage powder (both treatment & placebo) will be distributed in zip lock plastic bags to the participants by a third party (a graduate student) not involved in the study thereby keeping the investigators blind.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sedentary, overweight (BMI 25-29.9) females, between the ages of 18 - 25 years. Men will need to be measured in a separate study as there are likely gender differences and as this is an undergraduate student project there is insufficient time to assess both.

Exclusion Criteria:

* Women who are; unhealthy, currently physically active, taking medications, have health conditions contraindicated participation in exercise, allergic to milk, pregnant, or breastfeeding will be excluded.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Measuring changes in Lean Mass over 8 weeks at different time points | 4 weeks & 8 weeks
  Body lean mass (%) will be measured using BodPod

SECONDARY OUTCOMES:
Fat Loss changes over 8 weeks at different time points | 4 weeks & 8 weeks
  Body fat loss (%) will be measured using BodPod

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Research Laboratory, Western University, London, Ontario, Canada